CLINICAL TRIAL: NCT04453501
Title: Interest of Azithromycin With or Without Hydroxychloroquine for the Treatment of COVID-19 Pneumonia : a Retrospective Observational Study
Brief Title: Anti Infective Agents Impact in COVID-19 Pneumonia
Acronym: AZITHROVID
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Other Study IDs: AZITHROVID; INDS (Registry Identifier: MR1811190620)
Record Dates: First submitted 2020-06-25; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: COVID; Pneumonia, Viral
Keywords: azithromycin; hydroxychloroquine; COVID-19; pneumonia; hospitalization
MeSH Terms: conditions — Pneumonia, Viral; COVID-19; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Azithromycin or non-azithromycin group: Patient who received during admission for a severe COVID-19 pneumonia, azithromycin +/-hydroxychloroquine or no azithromycin.
  Interventions: Drug: favorable outcome

INTERVENTIONS:
Drug: favorable outcome — Whether patient under such regimen had a favorable outcome (no transfer in intensive care unit or death)

SUMMARY:
During COVID-19 epidemic, hydroxychloroquine was proposed and authorized as a possible key agent in the treatment of COVID-19 hospitalized pneumonia, including in France. Gautret et al. proposed the combination regimen with azithromycin. However only one study reported the interest of azithromycin alone.

Retrospective study reporting the impact of the anti-infective agents used during the pandemic in a tertiary care hospital, using azithromycin with or without hydroxychloroquine.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18 years old
* hospitalized for a COVID-19 pneumonia documented by PCR or lung tomodensitometry,
* admitted outside an intensive care unit, in a medicine ward

Exclusion Criteria:

* patient opposed to data collected, or who could not consent because of a serious presentation of the pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted at Hopital Raymond Poincaré, Garches, France in a medical ward for a COVID-19 pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
Favorable outcome | Assessed within 7 days after admission
  After being admitted, patient was monitored whether he does not required to be transferred in ICU or died because of a severe COVID-19 pneumonia within 7 days. The outcome was purely clinical. If patient was discharged at home after admission and/or was transferred into a rehabilitation center he was considered as a favorable outcome independently of any biological marker.

SECONDARY OUTCOMES:
Risk factors 1 | Assessed at day 1
  Studying if biological abnormalities (lymphocyte count or CRP) at admission were associated with an unfavorable outcome
Risk factors 2 | Assessed at day 1
  Studying if comorbidities were associated with an unfavorable outcome
Interest of anti-infective agents | From date of inclusion until the date of first documented progression to ICU or date of death from any cause, whichever came first, assessed up to 2 months
  Studying whether any regimen was associated with a favorable outcome (including azithromycin)

CONTACTS AND LOCATIONS:
Locations (1):
- Benjamin Davido, Garches, France

IPD SHARING:
Plan to Share IPD: No